CLINICAL TRIAL: NCT05610657
Title: A Phase 1, Open-label, Single-dose, Pharmacokinetic Study of Mitapivat in Subjects With Moderate Hepatic Impairment Compared to Matched Healthy Control Subjects With Normal Hepatic Function
Brief Title: A Pharmacokinetic Study of Mitapivat in Participants With Moderate Hepatic Impairment Compared to Matched Healthy Control Participants With Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AG348-C-024
Record Dates: First submitted 2022-11-03; First posted 2022-11-09 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Moderate Hepatic Impairment
Keywords: AG-348; Healthy Volunteer; Hepatic Impairment; pharmacokinetic
MeSH Terms: interventions — mitapivat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mitapivat (Experimental): Mitapivat tablet as a single oral dose, under fasted conditions on Day 1 to compare participants with normal hepatic function to participants with moderate hepatic function (Child-Pugh [C-P] Score B, score of 7 to 9).
  Interventions: Drug: Mitapivat

INTERVENTIONS:
Drug: Mitapivat — Mitapivat tablets
  Other Names: AG-348; AG-348 sulfate hydrate; Mitapivat sulfate

SUMMARY:
The primary purpose of this study is to compare the pharmacokinetics (PK) of a single oral dose of mitapivat in participants with moderate hepatic impairment to that in matched healthy control participants with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

For all Participants-

* Age: between 18 and 65 years of age;
* Men and women of any race;
* Body mass index (BMI) between 18.0 and 34.0 kilograms per square meter (kg/m^2), inclusive with at least 50 kg of body weight;
* There should be no use of tobacco- or nicotine-containing products within 3 months prior to check-in until completion of the follow-up visit;
* Male participants must agree not to donate sperm from check-in until 90 days after completion of the follow-up visit;
* Females of childbearing potential will agree to use contraception;
* Able to comprehend the requirements of the study and willing to sign an informed consent form before any study related procedures are conducted and to abide by the study restrictions.

For Participants with Normal Hepatic Function-

* In good health, determined by no clinically significant (CS) findings, as determined by the investigator, from medical and surgical history, physical examination, 12-lead ECG, vital signs measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [e.g., suspicion of Gilbert's syndrome based on total and direct bilirubin] is not acceptable) at screening and check-in;
* Serum electrolytes (sodium, potassium, chloride, bicarbonate, magnesium, and calcium) within normal limits or if deemed not CS by the investigator judgment in the case of minor abnormalities;
* Matched to participants with moderate hepatic impairment in sex, age (±10 years), and BMI (±20%).

For Participants with Moderate Hepatic Impairment-

* Diagnosis of chronic (≥3 months prior to screening) and stable hepatic insufficiency (no acute episodes of illness or deterioration in hepatic function) as assessed by the investigator with a C-P classification score of 7 to 9 (moderate hepatic impairment). Evidence of liver disease should be corroborated by medical history;
* Have current, or a history of at least 1 physical sign consistent with a clinical diagnosis of liver cirrhosis;
* Other than hepatic insufficiency with features of cirrhosis, hepatic impairment participants are in good health and clinically stable based on:

  * stable hepatic function is defined as no recent [i.e., within the preceding 14 days] CS change in disease status according to the investigator's clinical judgment (e.g., no worsening of clinical signs of hepatic impairment, or no worsening of total bilirubin or prothrombin by more than 50%).
  * the investigator's assessment including medical history and surgical history review, a defined complete physical examination, 12-lead ECG, vital signs, and clinical laboratory evaluations (clinical chemistry [including liver function tests], hematology, urinalysis, coagulation tests, thyroid function tests).
* Abnormal laboratory values (hepatic and nonhepatic) must be clinically acceptable by the investigator (or designee);
* Participants who need concomitant medications that are not prohibited during this study must have a medication regimen considered to be stable by the investigator. (e.g., no new drugs or significant changes to dosage(s) within 2 weeks [or 5 half-lives, whichever is longer] prior to study drug administration on Day 1; no changes expected during study conduct). Concomitant medications must be reviewed and approved by the investigator and Labcorp medical monitor (or designee).
* Anemia secondary to hepatic disease will be acceptable if hemoglobin is ≥8 grams per deciliter (g/dL) and anemia symptoms are not CS;
* Participants must have a platelet count ≥35 × 10^9/L.

Exclusion Criteria:

For all Participants-

* Presence or history of any disorder that may prevent the successful completion of the study;
* Participant is pregnant or breastfeeding;
* Significant acute, new-onset illness (e.g., flu, gastroenteritis) within 2 weeks prior to dosing;
* Inability to swallow medication;
* Has a history of relevant drug and/or food allergies (i.e., allergy to study drug or excipients [microcrystalline cellulose, croscarmellose sodium, sodium stearyl fumarate, mannitol, magnesium stearate, and the Opadry Blue II film-coat [hypromellose, titanium dioxide, lactose monohydrate, triacetin, and FD&C Blue #2]);
* Surgical or medical history that, in the opinion of the investigator, may potentially interfere with study drug absorption, distribution, metabolism, and/or excretion. Participants who have undergone abdominal surgery or any other major surgical procedure within 6 months prior to screening, must not be enrolled; The investigator should be guided by evidence of any of the following:

  1. History of inflammatory bowel syndrome, gastritis, ulcers, gastrointestinal or rectal bleeding within the past 3 months.
  2. History of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection.
  3. History of pancreatic injury or pancreatitis in the past 6 months; indications of impaired pancreatic function/injury as indicated by CS abnormal lipase or amylase.
  4. History of urinary obstruction or difficulty in voiding in the past 3 months.
* History or a presence of any malignancy, with the exception of a malignancy that has been curatively treated and for which the Participant has displayed no evidence of disease within 12 months prior to screening. Current or history of hepatic carcinoma, hepatorenal syndrome, portacaval shunt surgery, or pleural effusion. Malignancy, including leukemia and lymphoma, within the last 5 years. Participants with localized, fully-treated carcinoma of the skin may be allowed with investigator (or designee) approval;
* Confirmed (e.g., 2 consecutive measurements) systolic blood pressure >150 or <90 millimeters of mercury (mmHg), diastolic blood pressure >100 or <50 mmHg, and pulse rate >100 or <40 beats per minute (bpm); (Note: Participants with vital signs outside the above ranges may be eligible if the investigator and Labcorp medical monitor deem the results are not CS.)
* Clinically significant cardiac history or presence of ECG findings as determined by the investigator at screening and check-in, including any of the following:

  1. Abnormal sinus rhythm (heart rate [HR] lower than 40 bpm and higher than 100 bpm)
  2. Risk factors for torsades de pointes (e.g., heart failure, cardiomyopathy, or family history of long QT syndrome)
  3. Sick sinus syndrome, second- or third-degree atrioventricular block myocardial infarction, pulmonary congestion, cardiac arrhythmia, prolonged QT interval, or conduction abnormalities.
  4. QT interval corrected for HR using Fridericia's formula (QTcF) >450 milliseconds (msec) (healthy male participants) or >470 msec (healthy female participants) or >480 msec for hepatically impaired participants; in the event a QTcF value is outside of the reference range, it will be confirmed by 2 repeat measurements, which will then be used to calculate a mean from the original value and the 2 repeat measurements.
  5. QRS interval >110 msec, confirmed by manual over read.
  6. PR interval <120 and >220 msec.
  7. Repeated or frequent syncope or vasovagal episodes.
  8. Hypertension, angina, bradycardia (if assessed as CS by the investigator), or severe peripheral arterial circulatory disorders.
  9. History of autonomic dysfunction.
* Has estimated glomerular filtration rate <60 mL/minute/1.73 m^2 using Cockcroft-Gault equation;
* Administration of a coronavirus disease 2019 vaccine in the past 14 days prior to dosing;
* Has a positive test for severe acute respiratory syndrome coronavirus 2; Note: Testing will be performed according to site procedures;
* Has an active infection requiring systemic antimicrobial therapy at any time during the screening period;
* Is currently enrolled in or has participated in another clinical study to receive any investigational or marketed product or placebo within 4 weeks (or 5 half-lives, whichever is longer) or longer as required by local regulations prior to check-in;
* History of alcohol abuse within 3 months prior to screening and/or alcohol consumption of >21 units per week for males and >14 units for females. One unit of alcohol equals 12 ounce [oz] (360 mL) beer, 1 1/2 oz (45 mL) liquor, or 5 oz (150 mL) wine;
* Positive urine, breath, or blood test for alcohol or positive urine drug screen at screening and/or check-in;
* Positive urine cotinine test screening and/or at check-in (smokers will be defined as any participant who reports current tobacco use and/or who has a positive urine cotinine test);
* History or suspicion of active substance use disorder prior to check-in (including, but not limited to: cannabinoids, amphetamines, methamphetamines, 3,4-methylenedioxy-N-methylamphetamine [ecstasy], opiates, methadone, oxycodone, phencyclidine, cocaine, cotinine, benzodiazepines, and barbiturates);
* Ingestion of poppy seed-, Seville orange-, or grapefruit-containing foods or beverages within 7 days prior to check-in and not willing to refrain from consumption of these foods or beverages throughout the study until completion of the follow-up visit;
* Alcohol consumption, starting 48 hours prior to check-in and continuing until completion of the follow-up visit;
* Consumption of caffeine- or xanthine-containing products within 48 hours before check-in until completion of the follow-up visit;
* Consumption of vegetables from the mustard green family (e.g., kale, broccoli, watercress, collard greens, kohlrabi, Brussel sprouts, and mustard greens), or charbroiled meat for 7 days prior to dosing until completion of the follow-up visit;
* Receipt of blood products within 2 months prior to check-in;
* Participant has donated (or lost) ≥ 400 mL of red blood cells within 2 months prior to screening, plasma within 2 weeks prior to screening, or platelets within 6 weeks prior to screening; Participant has planned donation of any blood products after screening until 3 months after the follow-up visit;
* Participants are required to refrain from strenuous exercise from 7 days before check-in until completion of the follow-up visit and will otherwise maintain their normal level of physical activity during this time (i.e., will not begin a new exercise program nor participate in any unusually strenuous physical exertion);
* Poor peripheral venous access;
* Participants who, in the opinion of the investigator (or designee), should not participate in this study;
* Positive hepatitis B surface antigen or human immunodeficiency virus 1 or 2 test.

For Participants with Normal Hepatic Function-

* Liver test results (alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, albumin, or total bilirubin) above the upper limit of normal and/or prolonged prothrombin time (results may be repeated once), at screening and check-in, unless deemed not CS approved by the investigator (or designee);
* Has a known history or presence of liver disease;
* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder (as determined by the investigator);
* Uses or intends to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including slow-release medications/products, any over-the-counter medications or herbal or nutritional supplements with the exception of vitamins, within 14 days (or 5 half-lives, whichever is longer) prior to check-in and until completion of the follow-up visit, unless deemed acceptable by the investigator (or designee);
* Has used any prescription medications (excluding hormone replacement therapy, oral, implantable, transdermal, injectable, or intrauterine contraceptives), including systemic antimicrobial therapies, within 30 days (or 5 half-lives, whichever is longer) before dosing or during the study (ie, through the follow-up visit);
* Positive hepatitis C antibody;
* History of diabetes mellitus.

For Participants with Hepatic Impairment-

* Participants receiving strong and moderate cytochrome P450 (CYP) 3A inhibitors that have not been stopped for ≥5 days or a time frame equivalent to 5 half-lives (whichever is longer), or strong and moderate CYP3A inducers that have not been stopped for ≥4 weeks or a time frame equivalent to 5 half-lives (whichever is longer), before administration of the study drug;
* Participants with Grade 2 or higher encephalopathy, as defined by the grading scale in the Food and Drug Administration (FDA) guidance on PK studies in participants;
* Participant has a portal systemic shunt;
* Participant demonstrates evidence of hepatorenal syndrome;
* Participant has required treatment for gastrointestinal bleeding within the 3 months prior to check-in (Participants demonstrating banding procedure within 1 month prior to check-in may be included at the discretion of the investigator [or designee]);
* Participant has required new medication or a change in dose for hepatic encephalopathy within 3 months prior to check-in, unless approved by the investigator (or designee);
* Participants who require paracentesis within 3 months prior to check-in or planned during the study;
* Clinical evidence of moderate to severe ascites;
* Any evidence of progressive liver disease (between screening and check-in) as indicated by liver transaminases, alkaline phosphatase, or gamma-glutamyl transferase, or a ≥50% worsening of serum bilirubin or prothrombin time.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve From Time 0 (Predose) to Extrapolated to Infinity Time (AUC∞) of Mitapivat | Pre-dose and at multiple timepoints post-dose up to Day 17
Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUC0-t) of Mitapivat | Pre-dose and at multiple timepoints post-dose up to Day 17
Maximum Plasma Concentration (Cmax) of Mitapivat | Pre-dose and at multiple timepoints post-dose up to Day 17

SECONDARY OUTCOMES:
Time to Reach Cmax (tmax) of Mitapivat | Pre-dose and at multiple timepoints post-dose up to Day 17
Terminal Elimination Half-life (t1/2) of Mitapivat | Pre-dose and at multiple timepoints post-dose up to Day 17
Apparent Total Clearance (CL/F) of Mitapivat | Pre-dose and at multiple timepoints post-dose up to Day 17
Apparent Volume of Distribution During the Terminal Phase (Vz/F) of Mitapivat | Pre-dose and at multiple timepoints post-dose up to Day 17
Fraction Unbound (fu) for Mitapivat in Plasma | Pre-dose and at multiple timepoints post-dose up to Day 11
Number of Participants With Adverse Events (AEs), AEs by Severity, and Relatedness to Study Treatment | Up to Day 17
Number of Participants With Abnormalities in Laboratory Evaluations, Based on Coagulation, Hematology, Clinical Chemistry and Urinalysis Test Results | Up to Day 12
Number of Participants With Changes in 12-lead Electrocardiogram (ECG) Parameters | Up to Day 12
Number of Participants With Changes in Vital Sign Measurements | Up to Day 12
Number of Participants With Changes in Physical Examination Findings | Up to Day 12

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Study Chair — Agios Pharmaceuticals, Inc.
Locations (3):
- United States (3):
  - Orange County Research Center (OCRC), Tustin, California
  - Clinical Pharmacology of Miami (CPMI), Miami, Florida
  - Orlando Clinical Research Center (OCRC), Orlando, Florida

IPD SHARING:
Plan to Share IPD: No